CLINICAL TRIAL: NCT02861326
Title: RELATIONSHIP BETWEEN INITIAL PROBING DEPTH AND CHANGES IN CLINICAL PARAMETERS FOLLOWING NON-SURGICAL PERIODONTAL TREATMENT IN CHRONIC PERIODONTITIS PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Meseli
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Periodontitis
Keywords: chronic periodontitis, dental scaling, periodontal pockets
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Pocket

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Other): Non-surgical periodontal treatment has performed to patients. Scaling and root planing were performed with Gracey curettes until the operator feels that root surface is clean, hard and smooth.
  Interventions: Device: Gracey Curettes

INTERVENTIONS:
Device: Gracey Curettes
  Other Names: Hu-Friedy, SG 5/6, 7/8, 11/12, 13/14, Hu-Friedy Ins. Co., USA

SUMMARY:
Aim: The aim of this study was to evaluate the relationship between initial probing depth (IPD) and changes in clinical parameters following non-surgical periodontal treatment (NPT) in chronic periodontitis patients.

Material and Methods: A total of 1672 periodontal pockets having 3 mm≤IPD≤9 mm in 15 chronic periodontitis patients were included. NPT consisting of oral hygiene instructions, scaling and root planing was applied in two sessions. Probing depth (PD), clinical attachment level, gingival recession (GR) were measured before and eight weeks after treatment. Pocket sites were grouped according to their IPD and root number of teeth as single- or multi-rooted.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy,
* Non-smoker,
* Chronic periodontitis diagnosed according to Armitage 1,
* Aged between 35 and 65,
* Not received any periodontal treatment within the last 3 months, • Have horizontal bone loss radiographically,
* Presence at least 20 natural teeth except third molars
* Consent to participate in the study.

Exclusion Criteria:

* Any systemic disease that might interfere with the prognosis of periodontal disease (i.e. diabetes mellitus, HIV infection),
* Smoking,
* Antibiotics, anti-inflammatory drugs or any other medication taken within the previous 6 months that may affect the outcome of the study,
* Any physical limitations or restrictions that might preclude normal oral hygiene procedures.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Probing Depth | 8 week
  Probing depth is defined as the distance from the free gingival margin to the bottom of the periodontal pocket.

SECONDARY OUTCOMES:
Clinical attachment level | 8 week
  Clinical attachment level is defined as the distance from the cementoenamel junction to the bottom of the periodontal pocket
Gingival recession | 8 week
  Gingival recession is defined as the distance from cementoenamel junction to free gingival margin.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No